CLINICAL TRIAL: NCT00903110
Title: Global Patient Registry to Monitor Long-term Safety and Effectiveness of Increlex® in Children and Adolescents With Severe Primary Insulin-like Growth Factor-1 Deficiency (SPIGFD).
Status: Recruiting | Type: Observational
Sponsor: Esteve Pharmaceuticals, S.A. (Industry)
Responsible Party: Sponsor
Other Study IDs: 2-79-52800-002; EUPAS7708 (Other: EU PAS Register)
Record Dates: First submitted 2009-04-30; First posted 2009-05-15 (Estimated); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: IGF1 Deficiency
MeSH Terms: conditions — Insulin-Like Growth Factor I Deficiency | interventions — mecasermin

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: None Retained — Study Design Time Perspective: Retrospective and Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Increlex® — Increlex® (mecasermin [rDNA origin] injection), 10 mg/ml solution for injection, 40-120mcg/kg BID or 0,04 to 0,12 mg/kg BID, as prescribed by physician

SUMMARY:
The Increlex® Global Registry is a descriptive, multicenter, observational, prospective, open-ended, non interventional, post-authorisation surveillance registry.

The main purpose of this global registry is to collect, analyse and report safety data during and up to at least 5 years after the end of treatment in children and adolescents receiving Increlex® therapy for SPIGFD according to the locally approved product information.

DETAILED DESCRIPTION:
This registry is a Post-Authorisation Safety Study called the Increlex® Global Registry which is intended primarily to monitor the safety of Increlex® therapy in children and adolescents with Severe Primary IGF-1 Deficiency and secondly to follow the effectiveness of this treatment. Patients who have already started Increlex® therapy before entering this registry may be included and data will be collected retrospectively.

The countries participating in this registry are Austria, France, Germany, Italy, Poland, Spain, Sweden, United Kingdom and the USA

ELIGIBILITY:
Inclusion Criteria:

* For US : patients starting or planning to start or currently receiving treatment with Increlex® therapy for severe primary IGF-1 deficiency as defined by the US Increlex® prescribing information or for growth hormone (GH) gene deletion who have developed neutralizing antibodies to GH.For EU : patients starting or planning to start or currently receiving treatment with Increlex® therapy according to the locally approved product information.
* Parents or legally authorized representatives if applicable must give signed informed consent before any registry-related activities are conducted. Assent from the subject should also be obtained as appropriate

Exclusion Criteria:

* Subject currently participating in an Increlex® clinical trial
* Subject currently participating in any clinical trial for growth retardation
* Patient with any contraindication to Increlex® or any condition subject to special warning as per the locally approved label
* For US patients, these include patients with hypersensitivity to the active substance or any of the excipients, patients with active or suspected neoplasia and patients with closed epiphyses.
* For EU patients: these include patients with hypersensitivity to the active substance or any of the excipients, patients with active or suspected neoplasia or any condition or medical history which increases the risk of benign or malignant neoplasia and patients with closed epiphyses

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children and adolescents with Growth Failure due to Severe Primary IGF-1 Deficiency
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2008-12-09 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of SAEs (including AESI of neoplasia) and all AEs, targeted AEs, deaths and withdrawals due to AEs. | During the treatment period up to 30 days after the last dose.
  Targeted AE includes hypersensitivity; scoliosis; immunogenicity (presence of antibodies if available); slipped capital femoral epiphysis, headache, otitis media, papilloedema, hypoglycaemia (suspected or documented - documented means blood level glucose < 50 mg/dL or 2.78 mmol/L), acromegalic facial changes, gynaecomastia, hearing loss, intracranial hypertension, lipohypertrophy at injection sites, sleep apnoea, tonsillar hypertrophy, cardiomegaly, oedema and myalgia.

SECONDARY OUTCOMES:
Incidence of SAEs (including AESI of neoplasia), targeted AEs, all AEs, deaths, withdrawals due to AEs, special situations and concomitant medications | Within 5 years post-treatment
  In the overall population, and in the subset of children and adolescents exposed to Increlex® for at least 3 cumulative years excluding interruptions.
Incidence of special situations and concomitant medications | During the treatment period an average of 5 years and within 5 years post-treatment
Changes in height Standard Deviation Score (SDS) | From baseline at least up to 5 years or until the final adult height is achieved.
Height velocity | From baseline at least up to 5 years or until the final adult height is achieved.
Bone age development | From baseline at least up to 5 years or until the final adult height is achieved
Body mass index (BMI) | From baseline at least up to 5 years or until the final adult height is achieved.
Pubertal stage | From baseline at least up to 5 years or until the final adult height is achieved.
Estimation of differences between predicted adult height (PAH) and final adult height (FAH) | From baseline at least up to 5 years or until the final adult height is achieved.
Modelisation to identify predictive factors of height SDS change | From baseline at least up to 5 years or until the final adult height is achieved.
Modelisation to identify predictive factors of Height velocity | From baseline at least up to 5 years or until the final adult height is achieved
Modelisation to identify predictive factors of FAH | From baseline at least up to 5 years or until the final adult height is achieved
Modelisation to identify predictive factors of pubertal (Tanner) stage | From baseline at least up to 5 years or until the final adult height is achieved
Modelisation to identify predictive factors of bone age development | From baseline at least up to 5 years or until the final adult height is achieved
Dose of Increlex® administrated | Periodically assessed during the study until treatment stop at least up to 5 years.
Duration of Increlex exposure | Periodically assessed during the study until treatment stop at least up to 5 years.
Description of effectiveness parameters height SDS according to average dose received and according to dose ranges (e.g. 4 dose ranges (≤50, ]50-80], ]80-110], > 110 μg/kg BID)). | Periodically assessed during the study until treatment stop at least up to 5 years.
  This analysis will support the description of the lowest effective dose
Description of effectiveness parameters height velocity according to average dose received and according to dose ranges (e.g. 4 dose ranges (≤50, ]50-80], ]80-110], > 110 μg/kg BID)). | Periodically assessed during the study until treatment stop at least up to 5 years.
  This analysis will support the description of the lowest effective dose
Biological assessment : baseline GH concentrations, IGF-1 levels, IGFBP-3 levels and binding proteins. | Throughout study at least up to 5 years.
Presence or absence of gene deletion/mutation | Throughout study at least up to 5 years.
  including: GH gene, IGF-1 gene, FGF, PTPN11, GHR, D3-GHR, STAT5b, ALS, SHOX, PAPPA2 and any other genetic tests performed.
Changes in QoL assessment using EQ-5D in participant aged 4 and over. | At baseline, at year one, at least up to 5 years, at Final Adult Height.
  The QoL will be assessed using the EQ-5D-Y paediatric questionnaire. The 5 domains and VAS will be described at each timepoint as well as the evolution from baseline.
Description of neoplasia (benign and malignant) and hypoglycaemia | Within the first 3 years after treatment start, between 3 and 5 years and over 5 years.

CONTACTS AND LOCATIONS:
Overall Officials: Global Program Clinical Lead, Study Director — Esteve
Locations (58):
- United States (7):
  - Children's Hospital of Orange County, Orange, California
  - University of Miami Leonard M Miller, Miami, Florida
  - University Of Miami Leonard M. Miller, Miami, Florida
  - D&H National Research Centers, Miami, Florida
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - UT Southwestern Medical Center, Dallas, Texas
  - Children's Health Specialty Center West Plano, Plano, Texas
- Salzkammergut-Klinik Vöcklabruck, Vöcklabruck, Austria
- France (13):
  - Hôpital Amiens-Picardie, Amiens
  - Centre Hospitalier de Blois, Blois
  - Hôpital Jean Verdier, Bondy
  - Hôpital Femme Mère-Enfant, Bron
  - Hôpital Estaing, Clermont-Ferrand
  - Hôpital Timone Enfants, Marseille
  - Hôpital Arnaud de Villeneuve, Montpellier
  - GHR Mulhouse Sud-Alsace, Mulhouse
  - Pole medical Bel'Air, Mulhouse
  - CHU Lenval, Nice
  - Hôpital Necker Enfants Malades, Paris
  - Hôpital Kremlin Bicetre, Paris
  - Hôpital des Enfants, Toulouse
- Hôpital de Cayenne, Cayenne, French Guiana
- Germany (5):
  - Universitätsklinikum Erlangen Kinder- und Jugendklinik, Erlangen
  - Universitätsklinikum Heidelberg Kinderheilkunde, Heidelberg
  - Universitätskliniken des Saarlandes Kinderklinik, Homburg
  - Klinikum der Otto von Guericke Universität, Magdeburg
  - Klinikum Oldenburg, Oldenburg
- Italy (10):
  - Diabetologia Pediatrica Azienda Ospedaliero-Universitaria, Ancona
  - Ospedale di Bolzano, Bolzano
  - Spedali Civili di Brescia, Brescia
  - Azienda ospedaliera universitaria Meyer, Florence
  - I.R.C.C.S. Giannina Gaslini, Genova
  - U.O. Pediatria e Neonatologia Ospedale di Macerata, Macerata
  - Azienda Ospedaliera Universitaria II, Naples
  - Azienda Ospedaliera-Universitaria di Parma, Parma
  - Azienda USL-IRCCS, Reggio Emilia
  - Ospedale Pediatrico Bambino Gesù, Roma
- Hôpital Pierre Zobda Quitman, Fort-de-France, Martinique
- Poland (6):
  - Samodzielny Publiczny Dzieciecy Szpital Kliniczny, Bialystok
  - Uniwersyteckie Centrum Kliniczne, Gdansk
  - Uniwersytecki Szpital Dziecięcy w Lublinie, Lublin
  - Szpital kliniczny im. Karola Jonschnera, Poznan
  - Kliniczny Szpital Wojewódzki, Rzeszów
  - Pomeranian Medical University, Szczecin
- Spain (6):
  - Hospital Univ Vall d'Hebrón, Barcelona
  - Hospital Parc Taulí de Sabadell, Barcelona
  - Hospital Sant Joan de Déu, Barcelona
  - Hospital Univ. de Cruces, Bilbao
  - Hospital Universitari Sant Joan de Reus, Reus
  - Hospital Universitario y Politécnico La Fe, Valencia
- Sweden (2):
  - Linköping University Hospital, Linköping
  - Karolinska Universitetssjukhuset, Stockholm
- United Kingdom (6):
  - Royal Belfast Hospital for Sick Children, Belfast
  - Birmingham Children's Hospital, Birmingham
  - Leeds General Infirmary, Leeds
  - The Royal London Hospital, London
  - Great Ormond Street Hospital, London
  - Royal Manchester Children's Hospital, Manchester

REFERENCES:
- [Derived] Ramon-Krauel M, Polak M, Maghnie M, Woelfle J, Sert C, Perrot V, Bang P. Near-Adult Height Outcomes in Patients Treated With rhIGF-1 for Severe Growth Failure: Real-World IGFD Registry Data. J Clin Endocrinol Metab. 2026 Jan 21;111(2):e500-e511. doi: 10.1210/clinem/dgaf390. PMID 40626687
- [Derived] Bang P, Polak M, Bossowski A, Maghnie M, Argente J, Ramon-Krauel M, Sert C, Perrot V, Mazain S, Woelfle J. Frequency and Predictive Factors of Hypoglycemia in Patients Treated With rhIGF-1: Data From the Eu-IGFD Registry. J Clin Endocrinol Metab. 2023 Dec 21;109(1):46-56. doi: 10.1210/clinem/dgad479. PMID 37579214
- [Derived] Bang P, Polak M, Perrot V, Sert C, Shaikh H, Woelfle J. Pubertal Timing and Growth Dynamics in Children With Severe Primary IGF-1 Deficiency: Results From the European Increlex(R) Growth Forum Database Registry. Front Endocrinol (Lausanne). 2022 Feb 18;13:812568. doi: 10.3389/fendo.2022.812568. eCollection 2022. PMID 35250870
- [Derived] Bang P, Woelfle J, Perrot V, Sert C, Polak M. Effectiveness and safety of rhIGF1 therapy in patients with or without Laron syndrome. Eur J Endocrinol. 2021 Feb;184(2):267-276. doi: 10.1530/EJE-20-0325. PMID 33434161